CLINICAL TRIAL: NCT04021706
Title: Effect of a Ghrelin Receptor Agonist on Muscle and Bone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Bess Dawson-Hughes, Director Bone Metabolism Lab and Professor of Medicine, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3035; 1R21AR074138-01A1 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Sarcopenia; Osteopenia
MeSH Terms: conditions — Sarcopenia; Bone Diseases, Metabolic | interventions — anamorelin; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: double blind randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- anamorelin (Active Comparator): one 100 mg tablet daily, taken one hour before breakfast
  Interventions: Drug: Anamorelin Hydrochloride
- microcrystaline cellulose (Placebo Comparator): one identical appearing tablet daily, taken one hour before breakfast
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anamorelin Hydrochloride — Ghrelin receptor agonist
  Arms: anamorelin
Drug: Placebo — placebo is a inert substance
  Other Names: microcrystalline cellulose
  Arms: microcrystaline cellulose

SUMMARY:
Adults with low muscle mass also usually have low bone mass, making them vulnerable to falls, fractures and other injuries. This project will determine the effectiveness of treatment with a ghrelin receptor agonist in improving short term indicators of muscle and bone health in adults with low bone and muscle mass. The results of this trial will inform the design of a larger, definitive randomized trial designed to establish efficacy.

DETAILED DESCRIPTION:
Adults with both osteopenia and sarcopenia (osteosarcopenia) have greater risk of falls and fractures than those with osteopenia or sarcopenia alone. Drugs are available to reduce fracture risk but currently exercise is the only effective strategy to combat muscle loss. Unfortunately, the majority of adults who start a self-monitored exercise program drop out after 6 months and other options are needed. Ghrelin receptor agonists have been under development to treat anorexia and weight loss in patients with cancer cachexia. The agonist anamorelin has significantly increased weight and lean tissue mass in these patients. Anamorelin mimics the hormone ghrelin which not only increases appetite, but also acts on the pituitary to increase pulsatile growth hormone (GH) secretion. Pulsatile GH stimulates the production of insulin-like growth factor 1 which is anabolic to both muscle and bone. GH levels decline with age and this is thought to contribute to the age-related muscle and bone losses in adults. The central hypothesis is that anamorelin will increase muscle mass, improve muscle function, and increase bone formation in adults with osteosarcopenia. To test this hypothesis, the investigators will conduct a randomized, double-blind, 2-armed, parallel-group intervention trial in 32 osteosarcopenic men and postmenopausal women age 50 and older. Participants will be randomized to anamorelin (100 mg per day) or placebo and treated for 12 months. The primary endpoint is change from baseline in muscle mass by D3-creatine dilution. Secondary endpoints are:appendicular lean tissue mass/ht2 (ALM/ht2) measured by dual-energy x-ray absorptiometry (DXA); the bone formation biomarker, amino-terminal propeptide (P1NP), total body lean mass by DXA. Exploratory outcomes are changes in isokinetic leg strength, grip strength, and muscle performance (Health ABC-Physical Performance Battery (HABC-PPB), serum IGF-1 and C-telopeptide (CTX), and spine and hip bone mineral density (BMD). The proposed treatment supplies the anabolic stimulus to build both muscle and bone. Anamorelin has not been tested in adults with osteosarcopenia. The investigators propose to evaluate this treatment in osteosarcopenic adults who are most in need of treatment and who are also most likely to benefit. Data obtained from this pilot study are critical to determine the feasibility and guide the design of a definitive trial to evaluate this ghrelin receptor agonist as potential therapy to mitigate the dual hazards of osteopenia and sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to sign informed consent form
2. Community dwelling individuals aged 50 years and older

   1. Men (who are sterile or agree to use contraception throughout the study)
   2. Postmenopausal women (no menses for 5 years; early postmenopausal women are ineligible because their bone turnover rate is changing rapidly)
3. Sarcopenia defined as maximum grip strength <35.5 kg (men) and <20 kg (women) in either hand (excluding hands with severe pain or recent surgery) and/or gait speed <0.8 m/sec
4. Osteopenia defined as spine (at L1, L2, L3, or L4) or total hip or femoral neck BMD T-score between -1.0 and -2.5
5. Mini-mental state examination (MMSE) score >21

Exclusion Criteria:

1. BMI > 30 kg/m2 (obese are ineligible because anamorelin may cause weight gain)
2. Osteoporosis of the spine or hip by DXA scan (specifically, T-score ≤ -2.5 at two lumbar vertebrae or at the total hip or femoral neck, as recommended by the International Society for Clinical Densitometry [ISCD])
3. Current participation in a fitness program or weight loss program
4. Advanced knee osteoarthritis (OA) or other conditions preventing strength or function testing
5. Lower extremity fracture in the last year
6. Diabetics taking insulin or sulfonylureas and subjects with a fasting blood sugar on screening >150 mg/dl
7. Inadequate hepatic function defined as AST and ALT levels > 2 x upper limit of normal at screening (>74 and >68 MU/ml, respectively)
8. Untreated thyroid or parathyroid disease
9. Significant immune disorder
10. eGFR<30 ml/min
11. Any clinically meaningful electrocardiogram (ECG) abnormality on screening or baseline
12. Crohn's disease
13. Active malignancy or cancer therapy in the last year
14. Non-English speaking subjects (the investigators can't be confident that non-English speaking subjects could accurately complete the diet assessments which are critical to the integrity of the study)
15. Allergy to components of the study interventions
16. Other condition or abnormality in screening labs at discretion of the study physician (the PI)
17. Medications:

    1. Osteoporosis treatment - teriparatide, abaloparatide, raloxifene, denosumab, or romosozumab in the last 12 mo or a bisphosphonate in the last 2 years
    2. Tamoxifen in the last 6 mo
    3. Cancer treatment in the last 3 years (except basal cell skin cancer)
    4. strong CYP3A4 inhibitors within the previous two weeks (ketoconazole, clarithromycin, itraconazole, nefazodone, telithromycin)since anamorelin is mainly metabolized by CYP3A4
    5. Use of drugs that may prolong the PR or QRS interval durations, such as any of the Class I/Sodium (Na+) Channel blocking antiarrhythmic medications (e.g. flecainide, procainamide, propafenone, quinidine)
    6. Drugs with high affinity to alpha-acid glycoprotein (AAG) and therefore with potential to displace anamorelin from binding (e.g., carvedilol, chlorpromazine)
    7. Inhibitors of P-glycoprotein (e.g., verapamil, quinidine), and inhibitors of OATP1B3 (e.g., cyclosporine, rifampicin)
    8. CYP3A4 inducers (e.g., rifampin)
    9. Oral or IV glucocorticoids (>10 days in the last 3 mo)
    10. Gonadal hormones (vaginal estrogen okay)
    11. Drugs to promote weight loss or gain
    12. TNF-α inhibitors (e.g., adalimumab, adalimumab-atto, certolizumab pegol, etanercept, etanercept-szzs, golimumab, infliximab)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, MD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anamorelin | Microcrystaline Cellulose
Started | 17 | 15
Completed | 13 | 13
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are based on completers, 13 in each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anamorelin | Microcrystaline Cellulose | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (5.8) | 75.7 (6.4) | 74.5 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 11 | 11 | 22
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Total Body Muscle Mass
Description: to be assessed by D3-creatine dilution
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: kg units on a scale
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
kg units on a scale
  Baseline | 21.8 (4.8) | 20.8 (6.0)
  12 month visit | 22.2 (5.6) | 20.8 (7.4)

2. Secondary Outcome: Serum Procollagen 1 Intact N-terminal (P1NP)
Description: a serum biomarker of bone formation
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: micrograms/L
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
micrograms/L
  baseline | 42.0 (16.5) | 45.9 (33.7)
  12 month visit | 74.1 (45.4) | 46.2 (31.9)

3. Secondary Outcome: Fasting Plasma Glucose
Description: to be assessed by fasting blood drawn after 12 hour fast
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
mg/dL
  baseline | 95 (8.0) | 100 (8.0)
  12 month visit | 102 (16) | 97 (8.0)

4. Secondary Outcome: Serum Aspartate Transaminase (AST)
Description: to be assessed by blood drawn after 12 hour fast
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
U/L
  baseline | 23.2 (9.6) | 17.9 (3.8)
  12 month visit | 21.8 (8.4) | 17.8 (3.7)

5. Secondary Outcome: Alanine Transaminase (ALT)
Description: to be assessed by blood drawn after 12 hour fast
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
U/L
  baseline | 16.8 (6.9) | 17.8 (7.9)
  12 month visit | 15.8 (5.9) | 15.9 (6.3)

6. Secondary Outcome: Number of Participants With Symptoms and Any Adverse Events
Description: Number of participants with symptoms and any adverse events
Time Frame: between baseline and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
Participants
  Myalgia | 1 | 0
  Mild GI complaints | 2 | 0

7. Secondary Outcome: Appendicular Lean Mass (ALM)
Description: Dual energy X-ray absorptiometry (DXA) lean mass of arms plus legs
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
kg
  baseline | 20.8 (4.4) | 18.3 (3.8)
  12 month visit | 20.8 (4.4) | 18.0 (4.0)

8. Other Pre Specified Outcome: Handgrip Strength
Description: measure muscle strength and performance using grip strength dynamometer
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
kg
  baseline | 28.1 (8.3) | 25.0 (6.7)
  12 month visit | 28.4 (8.4) | 26.3 (7.3)

9. Other Pre Specified Outcome: Isokinetic Leg Strength
Description: measure muscle strength and performance using Biodex Isokinetic Dynamometer
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
Nm
  knee flexion at 240 degrees/sec - baseline | 27.5 (11.4) | 27.2 (9.0)
  knee flexion at 240 degrees/s, 12 month visit | 34.0 (11.2) | 27.8 (8.2)
  knee extension at 240 degrees/sec - baseline | 61.0 (18.5) | 56.1 (18.6)
  knee extension at 240 degrees/sec, 12 month visit | 65.2 (18.9) | 55.9 (18.1)

10. Other Pre Specified Outcome: Health Aging and Body Composition-Physical Performance Battery
Description: lower extremity performance score, scale from 0 (worst performance) to 4 (best performance)
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: score on a scale of 0 to 4
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
score on a scale of 0 to 4
  baseline | 2.25 (0.4) | 2.22 (0.4)
  12 month visit | 2.43 (0.4) | 2.35 (0.5)

11. Other Pre Specified Outcome: Serum Insulin Like Growth Factor-1 (IGF-1)
Description: anabolic intermediary of growth hormone
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
ng/mL
  baseline | 108 (14) | 110 (22)
  12 month visit | 162 (47) | 107 (38)

12. Other Pre Specified Outcome: Serum C-telopeptide (CTX)
Description: bone resorption marker
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
ng/mL
  baseline | 0.69 (0.2) | 0.72 (0.3)
  12 month visit | 0.73 (0.3) | 0.64 (0.3)

13. Other Pre Specified Outcome: Bone Mineral Density of the Spine and Hip
Description: assessed by DXA
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Anamorelin | Microcrystaline Cellulose
Number analyzed (Participants) | 13 | 13
g/cm^2
  Spine BMD at baseline | 1.03 (0.16) | 1.08 (0.17)
  Spine BMD at 12 months | 1.04 (0.16) | 1.09 (0.17)
  Femoral neck BMD at baseline | 0.73 (0.06) | 0.73 (0.08)
  Femoral neck BMD at 12 months | 0.72 (0.06) | 0.71 (0.07)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Anamorelin | Microcrystaline Cellulose
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/15
Other Adverse Events (participants affected / at risk) | 3/17 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin (N=17) | Microcrystaline Cellulose (N=15)
hematuria (Renal and urinary disorders) | 1 (2) | 0 (0) — hematuria
heart valve regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anamorelin (N=17) | Microcrystaline Cellulose (N=15)
GI bloating (Gastrointestinal disorders) | 2 (2) | 0 (0) — bloating
leaky heart valve (Cardiac disorders) | 0 (0) | 1 (1)
high blood sugar (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT04021706/Prot_SAP_000.pdf